CLINICAL TRIAL: NCT04386551
Title: Evaluation of the Performance of a Saliva Sample Versus a Nasopharyngeal Sample in the Diagnosis of COVID-19 by RT-PCR
Brief Title: Detection of COVID-19 in Saliva Collection
Acronym: SALICOV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0045
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Sars-CoV2; RT-PCR; Saliva Collection; Nasopharyngeal Sample
Keywords: Sars-CoV2; RT-PCR; Saliva collection; nasopharyngeal sample

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasopharyngeal sample and saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since December 2019, the world has faced a pandemic of COVID-19, an infectious disease caused by SARS-CoV-2, a virus that emerged in China. The reference diagnosis is based on the search for the SARS-COV-2 genome in the nasopharyngeal sample.

Carrying out this sample requires the competence of a healthcare professional and presents some inconveniences for the tested patient. Because saliva collection is simple, non-invasive, painless and inexpensive, and can be performed by poorly trained personnel, it could be an alternative to the reference nasopharyngeal sample. SARS-CoV2 detection in human saliva could be a potential diagnosis of COVID infection.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized at the Amiens CHU in a COVID-19 unit
* patient seen as outpatient in the area of infectious pathologies for COVID-19 infection

Exclusion Criteria:

* Patients under 18
* patients under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ambulatory patients screened for SARS Cov 19 at the CHU Amiens COViD clinic will be included in the study. A double sample will be taken from the saliva and the nasopharynx in parallel using the same sample kit. This double sampling has no direct impact on conventional patient management.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Detection of SARS-CoV-2 RNA in the saliva sample | day 1
  Detection of SARS-CoV-2 RNA in the saliva sample
Concordance between the Saliva sample and the nasonasopharyngeal sample SARS-CoV-2 RT-PCR results | day 1
  Concordance between the Saliva sample and the nasonasopharyngeal sample SARS-CoV-2 RT-PCR results

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No